CLINICAL TRIAL: NCT00248378
Title: Short-Term Effects of Medicinal Cannabis Therapy on Spasticity in Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Center for Medicinal Cannabis Research (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: C00-SD-103; 030002
Record Dates: First submitted 2005-11-02; First posted 2005-11-04 (Estimated); Last update posted 2006-06-23 (Estimated); Status verified 2006-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Cannabis; Spasticity; Tolerability
MeSH Terms: conditions — Multiple Sclerosis; Marijuana Abuse; Muscle Spasticity

INTERVENTIONS:
Drug: Smoked Cannabis

SUMMARY:
The purpose of this study is to determine whether or not smoked marijuana improves spasticity in patients with multiple sclerosis.

DETAILED DESCRIPTION:
Studies of cannabinoids for spasticity in MS have had mixed results but clinical studies have been small, generally not properly controlled, with results controversial, and difficult to interpret. Recently, investigators in the UK and US tested the ability of cannabinoids to control spasticity and tremor symptoms of the MS-like disease, experimental allergic encephalomyelitis, in mice (Baker et al, 2000). The authors found that four different cannabinoids quantitatively ameliorated both tremor and spasticity in diseased mice; thus providing rationale for patients' reports of the therapeutic effects of cannabis in the control of their MS symptoms.

The present study will be a randomized, placebo-controlled, crossover design of 30 patients who will be assessed before and after treatment for 3 consecutive days (Phase I), undergo washout-out for a total of 11 days, and then cross over to either the placebo or active treatment phase (Phase II), depending on what they received during Phase I. At each study visit, patients will utilize a controlled puff procedure to help ensure stable intake (Levin et al, 1989).

Comparisons: A single dose of 4% THC marijuana cigarette each day for 3 days will be compared to a placebo administered under the same dosing conditions for the relief of spasticity, drug tolerability, and changes in global functioning and quality of life indices.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite or probable, laboratory-supported MS
* Complaints of spasticity and at least moderate increase in tone as evidenced by a score of >= 2 on the Modified Ashworth Scale at either the elbow, hip, or knee
* If on disease-modifying therapy ("ABC"), have been on a stable dose for at least six months
* Fluent in English
* If not cannabis-naive, must refrain from smoking cannabis for two weeks prior to screening (confirmed by urinalysis)
* If on either lioresal (Baclofen) or tizanadine (Zanaflex), have been on a stable dose for at least three months
* >=18 years of age

Exclusion Criteria:

* Axis I psychiatric disorder especially depression or significant neurological disease other than MS as determined by the PI
* Recent history of active substance abuse defined as daily use for at least 14 days within the past month
* Drug use restrictions, eg, subjects on probation or parole, employment involving high risk to themselves and/or the public (airline pilot, bus driver, etc.)
* Any unstable medical health problem
* Any known pulmonary disorders, including tuberculosis, asthma, or COPD
* Pregnant or nursing
* Require benzodiazepines to control spasticity
* Require high doses of analgesic medications on a daily basis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2001-09; Study Completion 2005-03

PRIMARY OUTCOMES:
Reduction in spasticity as indicated by the: Ashworth Spasticity Scale, Timed 25-ft Walk, and Grooved Pegboard Test

SECONDARY OUTCOMES:
Tolerability of study drug as determined by the Brief Symptom Inventory, Subjective Ratings of High and Sedation-Revised, and UKU Side Effect Rating Scale
Effect of study drug on global functioning and quality of life as indicated by the Multiple Sclerosis Quality of Life Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Jody Corey-Bloom, M.D., Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego Medical Center, San Diego, California, United States

REFERENCES:
- See also: Center for Medicinal Cannabis Research — http://cmcr.ucsd.edu